CLINICAL TRIAL: NCT02361385
Title: Pilot Study to Evaluate the Feasibility of [11C]PBR28 PET-CT to Image Inflammation in the Joints of Arthritis Patients
Brief Title: PBR28 PET and Inflammatory Arthritis
Status: Completed | Type: Observational
Sponsor: University of Oxford (Other)
Collaborators: Imanova Centre for Imaging Sciences (Unknown)
Responsible Party: Sponsor
Other Study IDs: 11132
Record Dates: First submitted 2015-02-06; First posted 2015-02-11 (Estimated); Last update posted 2018-10-12 (Actual); Status verified 2018-05

CONDITIONS: Rheumatoid Arthritis; Psoriatic Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid; Arthritis, Psoriatic

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — A single blood sample will be taken for a genotyping test, to ascertain whether or not individuals are suitable to undergo PET-CT with the PBR28 PET tracer. Further, blood samples will be taken for serum and RNA, and synovial biopsy will be done.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- this is a pilot study: All patients will undergo PET-CT with PBR28, with the CT being localised to one group of joints only
  Interventions: Other: this is not an interventional study

INTERVENTIONS:
Other: this is not an interventional study — this is not an interventional study; this is a pilot feasibility study to see whether or not 11CPR28 will be taken up in joints of those known to have active arthritis clinically

SUMMARY:
The importance of the detection of early inflammatory arthritis is recognised as being essential to the prevention of permanent joint damage. Furthermore, drug development in inflammatory arthritis is in increasing need of imaging that is able to sensitively and accurately detect and quantify inflammation in a reproducible and objective manner. There is an increasing body of evidence to support the role of PET-CT for these indications. The PET tracer 11CPBR28 is specific to the translocator protein (TSPO) highly expressed on activated macrophages. In this proof of principle study, the investigators aim to ascertain whether or not the PET tracer 11CPBR28 is taken up in inflamed joints. The investigators also aim to explore the significance of TSPO to inflammatory arthritis, through blood and joint lining samples.

DETAILED DESCRIPTION:
The investigators aim to recruit a minimum of 12 patients with known, active rheumatoid or psoriatic arthritis in the feet and ankles. Patients will first undergo a screening genotyping test; low affinity binders for PBR28 PET will be excluded from this pilot study. Those patients meeting inclusion criteria, will then undergo a PET-CT localised to feet and ankles that have been identified to be clinically inflamed (on examination and ultrasound at the screening visit). After PET-CT, patients will undergo synovial biopsy of one joint imaged. After 6 patients have undergone PET-CT, an interim analysis will be undertaken, to optimise PET scan duration and to alter the group of joints being imaged with CT.

ELIGIBILITY:
Inclusion Criteria:

* Patients with known rheumatoid arthritis or psoriatic arthritis, with at least one swollen joint, with evidence of joint inflammation in the feet and/or ankles (on clinical examination and/or ultrasound)

Exclusion Criteria:

* pregnant and breastfeeding patients those with metalwork in feet/ankles patients unable to lie on their back Patient has been identified as a low affinity [11C]PBR28 binder according to peripheral blood genotyping assay The patient has any significant co-morbidity precluding participation as judged by the study doctor

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with known rheumatoid arthritis or psoriatic arthritis, with at least one swollen joint, with evidence of joint inflammation in the feet and/or ankles (on clinical examination and/or ultrasound)
Sampling Method: Non-Probability Sample
Enrollment: 22 (Actual)
Dates: Start 2015-03 (Actual); Primary Completion 2017-07 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
standardised uptake values (SUV) | maximum duration of scan is 90 minutes
  Evidence of uptake of 11CPBR28 in the inflamed feet and/or ankle joints of patients with known rheumatoid or psoriatic arthritis as exhibited by SUV (standard uptake values) on the PET-CT images.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Taylor, MA,BChB,FRCP, Principal Investigator — University of Oxford
Locations (2):
- United Kingdom (2):
  - Imanova Centre for Imaging Sciences, London, Greater London
  - Nuffield Orthopaedic Centre, Oxford, Oxfordshire